CLINICAL TRIAL: NCT04340700
Title: Characterization of the Pharmacodynamic Response to Vaped THC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding not received
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director, Center for Addiction Medicine; Professor in Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2020P000055
Record Dates: First submitted 2020-03-23; First posted 2020-04-09 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Vaping; THC
Keywords: Vaping; THC; fNIRS; Cannabis; Imaging
MeSH Terms: conditions — Vaping; Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- THC (Experimental): A standard dose of THC (8 mg or 2 mg) will be placed in a Volcano Vaporizer chamber. The first THC dose is 8 mg, followed by approximately three doses of 2 mg each.
  Interventions: Drug: THC or Placebo
- Placebo (Placebo Comparator): Placebo will also be administered through a Volcano Vaporizer via inhalation. The first placebo dose is 8 mg, followed by approximately three doses of 2 mg each to match the THC procedures.
  Interventions: Drug: THC or Placebo

INTERVENTIONS:
Drug: THC or Placebo — A standard dose of THC (8 mg or 2 mg) will be placed in a Volcano Vaporizer chamber. The first THC dose is 8 mg, followed by approximately three doses of 2 mg each. Placebo will also be administered through a Volcano Vaporizer via inhalation. The first placebo dose is 8 mg, followed by approximately three doses of 2 mg each to match the THC procedures.

SUMMARY:
This study aims to characterize the pharmacodynamic response to vaped THC in young adult, occasional cannabis users with respect to outcomes such as stimulation and sedative effects, mood, anxiety, and craving, as well as cognitive and objective outcomes such as heart rate and cortisol changes with THC vs placebo.

DETAILED DESCRIPTION:
Enrollees will include 120 healthy, weekly or greater MJ users, aged 18-55. The study will be conducted according to a double-blind, placebo-controlled, random order, cross-over design, consisting of one 3-hour screening visit and 2 randomized, approximately 6-hour laboratory sessions. At the latter visits (following confirmation of eligibility), subjects will complete baseline questionnaires and assessments, including a driver simulator test, a blood draw, vitals, and an imaging session using functional near-infrared spectroscopy (fNIRS). Subjects will then vape a first dose (either THC or placebo based on randomization). Vitals and questionnaires will then be administered throughout the visit, at baseline, and at approximately 15, 60, 90, 130, 165, and 210 minutes post initial dose. Subjects will also perform fNIRS testing at baseline, 30, and 180 minutes and driver simulator at baseline, 60, and 90 minutes post initial THC/placebo administration. A drug recognition expert (DRE) will conduct a standard field sobriety test to identify impairment at approximately 130 minutes post dose. Following the initial dose vaped at 0 minutes, standardized reduced doses will be vaped approximately 30, 60, and 90 minutes later. Given the cross-over design of this study, participants will be assigned to receive THC or placebo at the first laboratory visit and will receive the other substance at the second laboratory visit.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-55 years, inclusive.
* Competent and willing to provide written informed consent.
* Able to communicate in English language.
* Regular, at least weekly on average, marijuana use
* Self-reported ability to abstain from cannabis for 24 hours without withdrawal.

Exclusion Criteria:

* Any unstable, serious medical illness or cardiovascular disease/events.
* New or unstable psychiatric symptoms, schizophrenia, or bipolar I disorder.
* Diabetes, cirrhosis, renal failure, Hepatitis C, or HIV.
* History of syncope without an identified situational stressor, migraines >1x/month, or head injury with prolonged unconsciousness (> 24 hours).
* Daily use of benzodiazepines or barbiturates, antihistamines, atropine, scopolamine, or other strong anticholinergic agents.
* Current pregnancy, lactation or trying to become pregnant (confirmed by urine pregnancy test).
* History of substance abuse treatment and intent to quit or receiving treatment for cannabis use.
* Affective disorder in the past month or history of panic attacks.
* Smoking more than 10 tobacco cigarettes or equivalent e-cigarettes a day.
* In the opinion of the investigator, not able to safely participate in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Drug Effects Questionnaire | Pre-dose, and 15, 60, 90, 130, 165, 210 minutes post dose
  This 15-item questionnaire measures drug effects, behavioral/mood states, and craving. Each item is scored from 0-100, and all items are averaged for a total score from 0-100 with higher scores indicating greater drug effect.
Change in Biphasic Alcohol Effects Scale (Modified for THC) | Pre-dose, and 15, 60, 90, 130, 165, 210 minutes post dose
  This 14-item questionnaire measures stimulation and sedation. The Stimulation subscale scores range from 7-70 with higher scores indicating greater stimulation. The Sedation subscale scores range from 7-70 with higher scores indicating greater sedation.
Change in The Spielberger State Anxiety Inventory | Pre-dose, and 15, 60, 90, 130, 165, 210 minutes post dose
  This 20-item questionnaire measures state/current anxiety. Scores range from 20-80 with higher scores indicating greater state anxiety.
Change in Driving Simulation Performance on the Divided Attention Task (DAT) | Pre-dose, and 60 and 90 minutes post dose
  A computer-programmed driving simulator will assess DAT performance using percentage impaired (from 0-100%).

SECONDARY OUTCOMES:
Change in Functional Near-Infrared Spectroscopy (fNIRS) Brain Signal | Pre-dose, and 30 and 180 minutes post dose
  fNIRS measures oxygenated hemoglobin (HbO) during both resting state and a working memory task in both THC and placebo conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No